CLINICAL TRIAL: NCT01653106
Title: A Randomized Study to Compare the Effect of Short- and Long-Term Schedules of Cryotherapy on the Incidence and Severity of Mucositis in High-Dose Melphalan
Brief Title: Randomized Trial of Cryotherapy Duration Prior to High Dose Melphalan in Myeloma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Craig Hofmeister, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-11055; NCI-2012-00459 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
Keywords: cryotherapy; Melphalan; Mucositis
MeSH Terms: conditions — Multiple Myeloma; Mucositis | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cryotherapy 120 minutes) (Experimental): Beginning fifteen minutes before melphalan treatment, patients receive 1 ounce of shaved ice in their mouth, allow it to melt and then replenish it immediately for 120 minutes.
  Interventions: Procedure: cryotherapy; Other: questionnaire administration; Other: pharmacological study
- Arm II (cryotherapy 360 minutes) (Active Comparator): Beginning fifteen minutes before melphalan treatment, patients receive 1 ounce of shaved ice in their mouth, allow it to melt and then replenish it immediately for 360 minutes.
  Interventions: Procedure: cryotherapy; Other: questionnaire administration; Other: pharmacological study

INTERVENTIONS:
Procedure: cryotherapy — Receive shaved ice
Other: questionnaire administration — Participate in PROMS
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
The purpose of this study is to compare the effect of short-term (2 hours/120 minutes) and long-term (6 hours/360 minutes) schedules of crushed ice therapy (cryotherapy). Patients that receive high dose melphalan for bone marrow transplantation commonly develop significant mouth pain and sores (oral mucositis) unless cryotherapy is utilized. The goal of this study is to scientifically determine (using randomization and a larger sample size) if a short-term schedule is as effective as the standard long-term schedule in preventing, or minimizing the symptoms involved with oral mucositis. The study is also trying to determine the best dose of melphalan and how patient's body breaks down melphalan and will obtain blood through central venous catheter to measure the amount of melphalan in patient's blood at specific times after the melphalan is infused

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the maximum inpatient mucositis grade after 120- vs. 360-minutes standardized cryotherapy regimens in patients with multiple myeloma undergoing autologous hematopoietic stem cell transplantation at Ohio State Medical Center.

SECONDARY OBJECTIVES:

I. To develop a pharmacokinetic model predicting variability in unbound serum melphalan area under the concentration-time curve (AUC).

II. To compare the neutropenic fever and bacteremia incidence after 120- vs. 360-minute cryotherapy regimens.

III. To compare patient-reported mucositis-related symptoms up until discharge utilizing the Patient-Reported Oral Mucositis Symptoms Scale (PROMS) after 120- vs 360-minute cryotherapy regimens.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Beginning fifteen minutes before melphalan treatment, patients receive 1 ounce of shaved ice in their mouth, allow it to melt and then replenish it immediately for 120 minutes.

ARM II: Beginning fifteen minutes before melphalan treatment, patients receive 1 ounce of shaved ice in their mouth, allow it to melt and then replenish it immediately for 360 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with multiple myeloma be admitted for autologous stem cell transplantation
* Age > 18 years
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial

Exclusion Criteria:

* Any other medical condition, including mental illness or substance abuse, deemed by the principal investigator to likely interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of severe (Grade 3 or 4) mucositis achieved between two different cryotherapy regimens during inpatient hospitalization based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | 21 days
  A Cochran-Mantel-Haenszel chi-square test will be used to compare the proportion of patients who develop severe mucositis between those treated with 120-minute vs. 360-minute cryotherapy. Logistic regression modeling will also be used with incidence of severe mucositis as the dependent variable and assess various factors in addition to treatment arm on this incidence.

SECONDARY OUTCOMES:
Melphalan pharmacokinetic model including apparent volume of the central compartment (Vc), elimination rate of constant (Ke), half-life (t1/2), systemic clearance (CLs), and AUC. | Pre-dose, within 5 minutes prior to completion of infusion, at 5, 15, 30, 45, and 60 minutes, and 3 and 6 hours post end of infusion
  All pharmacokinetic results will be summarized using appropriate descriptive statistics. A nonlinear mixed effects approach will be used for modeling melphalan pharmacokinetics, identifying significant covariates, and relating these to mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Poi MJ, Li J, Sborov DW, VanGundy Z, Cho YK, Lamprecht M, Pichiorri F, Phelps MA, Hofmeister CC. Polymorphism in ANRIL is associated with relapse in patients with multiple myeloma after autologous stem cell transplant. Mol Carcinog. 2017 Jul;56(7):1722-1732. doi: 10.1002/mc.22626. Epub 2017 Feb 16. PMID 28150872
- See also: Jamesline — http://cancer.osu.edu